CLINICAL TRIAL: NCT00712738
Title: A Trial of Oral Nifedipine for the Treatment of Iron Overload
Brief Title: Oral Nifedipine to Treat Iron Overload
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Jeffery L. Miller, M.D./National Institute of Diabetes and Digestive and Kidney Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080157; 08-DK-0157
Record Dates: First submitted 2008-07-09; First posted 2008-07-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-09-22

CONDITIONS: Thalassemia; Iron Overload; Hemochromatosis
Keywords: Nifedipine; Thalassemia; Hemochromatosis; Iron Overload; Iron Excretion
MeSH Terms: conditions — Thalassemia; Iron Overload; Hemochromatosis | interventions — Nifedipine; Phlebotomy; Urinalysis

INTERVENTIONS:
Drug: Nifedipine
Procedure: Phlebotomy
Procedure: Urinalysis
Procedure: Echocardiogram
Procedure: Electrocardiogram

SUMMARY:
This study will determine if nifedipine, a medication used to treat high blood pressure, can help treat iron overload, a condition in which the body contains too much iron. Iron overload can be caused by the body's inability to regulate iron or by medical treatments, such as multiple blood transfusions. Over time, it can cause problems with the liver, heart and glands. Treatments include reducing iron intake in the diet or removing the excess iron using medical therapies. Recently, nifedipine was found to cause iron loss in the urine of small animals. This study will see if the drug can increase the removal of iron into the urine in humans as well.

People 18 years of age and older with iron overload may be eligible for this study to undergo the following procedures:

Study Day 1

Participants come to the NIH Clinical Center for a medical history, physical examination, blood and urine tests, electrocardiogram (EKG) and echocardiogram (heart ultrasound).

Study Day 2

Participants will collect three urine samples: one is collected over 4 hours, followed by a second over 4 hours. Both of these samples are collected at NIH in the outpatient day hospital. At home, a third urine sample will be collected over 16 hours. For 1 week before the collections, participants are asked not to drink tea or eat foods high in Vitamin C or iron. They are also asked not to take any iron chelating medications.

Study Day 3

Participants repeat the same urine collections as on day 2. They collect a 4-hour urine sample at the outpatient day hospital at NIH. They will then take a 20-mg tablet of nifedipine, and remain in the clinic 4 hours for blood pressure monitoring. A second urine sample during this time. They then return home to collect the final 16-hour sample, which they bring to the clinic the following day. Again, they are instructed to avoid a diet high in vitamin C, iron rich foods, tea, and to avoid taking any iron chelating medications.

...

DETAILED DESCRIPTION:
Iron overload is common worldwide. If left untreated, body iron overload leads to multiple organ abnormalities including hepatic, endocrine (diabetes) and cardiac failure. In patients with ineffective erythropoiesis, iron overload results from the combination of increased intestinal absorption and transfusion. Unfortunately, physiological means to remove excess iron are limited, and treatments are limited to therapeutic phlebotomy and chelation therapy. While phlebotomy is the preferred therapy for patients with hemochromatosis, therapy for anemic patients is largely limited to chelation drugs. Since those drugs are frequently inadequate, additional iron-reduction therapies are being sought. Based upon recently published data in a rodent model, the purpose of this study is to determine if nifedipine will increase iron excretion in the urine among humans with increased levels of iron. Volunteers will be given a single oral dose (20mg) of nifedipine. Iron level in collections of urine will be measured and compared before and after nifedipine to determine if there is an associated increase in urinary iron excretion.

ELIGIBILITY:
* INCLUSION CRITERIA:

Iron overloaded subjects will have a history of iron overload that may be due to a variety of causes including genetic hemochromatosis or thalassemia or other transfusion-dependent anemias (e.g. sickle cell syndromes, aplastic anemia, ineffective erythropoiesis) or other causes. Entry into the study requires that all subjects possess at least minimal evidence of iron overload at the time of entry (defined as serum ferritin and serum transferrin saturations levels above the normal range). Among fifty (50) subjects recruited for this protocol, at least twenty (20) with significant iron overload (defined in this study as ferritin greater than 500 ng/ml and transferrin saturation greater than (50%) will be included.

All subjects will be of adult age (greater than or equal to 18 yrs).

All subjects enrolled in this protocol will have a primary physician and care in the community that is capable of managing any medical problems unrelated to the nifedipine regimen.

All subjects must be able to provide informed consent.

EXCLUSION CRITERIA:

Allergy to nifedipine.

Patient receiving calcium channel blocker therapy within 7 days prior to enrollment.

Blood transfusion within 7 days of first urine iron evaluation.

Pregnant or lactating women.

Patients with GFR less than 60 ml/min.

Albumin less than 3g/dl.

Significant hemoglobinuria (greater than1+ on urinalysis).

Hemoglobin less than 10 g/dl

Uncompensated cardiac disease including decreased ejection fraction detected by echocardiogram, angina, hypotension (less than 90mmHg systolic pressure) or symptomatic arrhythmias. Documented myocardial infarction within one year prior to the study.

Use of tea, Vitamin C, iron chelation therapy, iron supplements, grapefruit juice, cimetidine, digitalis, quinidine, or beta-blockers (due to potential for increased serum drug levels versus cardiovascular risk) within 7 days prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-06-20; Primary Completion 2010-09-22 (Actual); Study Completion 2010-09-22 (Actual)

PRIMARY OUTCOMES:
Evaluate nifedipine-related urinary iron excretion.

SECONDARY OUTCOMES:
Evaluate potential for nifedipine to increase urinary iron excretion among patients with iron overload.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cappellini MD, Cohen A, Piga A, Bejaoui M, Perrotta S, Agaoglu L, Aydinok Y, Kattamis A, Kilinc Y, Porter J, Capra M, Galanello R, Fattoum S, Drelichman G, Magnano C, Verissimo M, Athanassiou-Metaxa M, Giardina P, Kourakli-Symeonidis A, Janka-Schaub G, Coates T, Vermylen C, Olivieri N, Thuret I, Opitz H, Ressayre-Djaffer C, Marks P, Alberti D. A phase 3 study of deferasirox (ICL670), a once-daily oral iron chelator, in patients with beta-thalassemia. Blood. 2006 May 1;107(9):3455-62. doi: 10.1182/blood-2005-08-3430. Epub 2005 Dec 13. PMID 16352812
- [Background] Barton JC. Chelation therapy for iron overload. Curr Gastroenterol Rep. 2007 Mar;9(1):74-82. doi: 10.1007/s11894-008-0024-9. PMID 17335681
- [Background] Ludwiczek S, Theurl I, Muckenthaler MU, Jakab M, Mair SM, Theurl M, Kiss J, Paulmichl M, Hentze MW, Ritter M, Weiss G. Ca2+ channel blockers reverse iron overload by a new mechanism via divalent metal transporter-1. Nat Med. 2007 Apr;13(4):448-54. doi: 10.1038/nm1542. Epub 2007 Feb 11. PMID 17293870
- [Derived] Padhani ZA, Gangwani MK, Sadaf A, Hasan B, Colan S, Alvi N, Das JK. Calcium channel blockers for preventing cardiomyopathy due to iron overload in people with transfusion-dependent beta thalassaemia. Cochrane Database Syst Rev. 2023 Nov 17;11(11):CD011626. doi: 10.1002/14651858.CD011626.pub3. PMID 37975597